CLINICAL TRIAL: NCT00631332
Title: Effects of Hormone Replacement Therapy on Cognitive Aging: Women's Health Initiative Study of Cognitive Aging (WHISCA)
Brief Title: Women's Health Initiative Study of Cognitive Aging
Acronym: WHISCA
Status: Completed | Type: Observational
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Other Study IDs: NO1-AG-9-2115
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-06

CONDITIONS: Healthy
Keywords: women, dementia, cognition.; non-demented women at least age 65
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Women's Health Initiative Study of Cognitive Aging (WHISCA) is a two-armed, randomized, placebo controlled, clinical trial designed to assess the efficacy of postmenopausal hormone therapy (HT) on age related changes in specific cognitive functions.

DETAILED DESCRIPTION:
WHISCA is an ancillary study to the Women's Health Initiative (WHI) and the WHI Memory Study (WHIMS) and has enrolled 2303 women aged 66 to 84 years who did not meet the criteria for dementia. WHISCA is investigating the effects of hormone therapy on rates of change over time in memory, other aspects of cognition (language, attention, spatial ability), motor function, and mood.

Objectives

* Does HT protect against age-associated memory and cognitive longitudinal decline in women age 65 and older?
* What is the rate of change in memory and other cognitive abilities in women receiving HT compared to women receiving placebo?
* Does the addition of progesterone to HT modify the effects of estrogen on memory and other cognitive abilities?

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in WHIMS
* At least 65 years old
* Not diagnosed with dementia

Exclusion Criteria:

* Women younger than 65 years of age
* Have dementia
* not enrolled in WHIMS

Ages: 65 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: A subset of women who were enrolled in the Women's Health Initiative Memory Study (WHIMS), who are at least 65 years old and not diagnosed with any type of dementia.
Sampling Method: Non-Probability Sample
Enrollment: 2303 (Actual)
Dates: Start 1999-07; Primary Completion 2007-09 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Determine if HT protect against age-associated memory and cognitive longitudinal decline in women age 65 and older as measured over time by a series of cognitive tests administered annually. | Annual assessment done annually.
  The primary outcome measures are the changes in scores from a standardized neuropsychological assessment will be conducted annually. The battery is comprised primarily of tests of memory, and includes the following tests in specified order: the Prospective Memory Tests, Primary Mental Abilities Vocabulary Test, the California Verbal Learning Test, the Benton Visual Retention Test, Card Rotations Test, the Finger Tapping Test, the Letter and Semantic Fluency Test and the Digit Span Test. In addition, the Positive and Negative Affect Scale and Geriatric Depression Scale will be administered.

SECONDARY OUTCOMES:
Determine the long-term effects of HT on changes in memory, other cognitive functions, and affect; and to investigate predictors of the transitions between normal aging and mild cognitive impairment and mild cognitive impairment and dementia. | measured over life of the study
  Secondary outcome measures will examine relative differences in measures between enrollment in WHIMS and the termination of the WHIMS E+P trial and E-Alone trial and also examine the relative differences in measures comparing periods of time for each woman when she reported taking HT versus times she reported not taking HT.

CONTACTS AND LOCATIONS:
Overall Officials: Sally Shumaker, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University School of Medicine, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
WHISCA will follow guidelines, methods and processes as set forth in the WHI 2015-2020 Data Sharing Plan. Accompanying the limited data sets, substantial electronic documentation will be provided in a standard format that is readable on a variety of platforms. Documentation will include data collection forms, a description of study protocol and procedures, description of all variable re-coding and a list of major study publications. These data will be available to users only under a data-sharing agreement that provides for: a commitment to using the data only for research purposes and not to identify any individual participant; a commitment to securing the data using appropriate computer technology; and a commitment to destroying or returning the data after analyses are completed. Data will be made available for timely release no later than the acceptance for publication of the main findings from the final dataset.

REFERENCES:
- [Background] Ammann EM, Pottala JV, Harris WS, Espeland MA, Wallace R, Denburg NL, Carnahan RM, Robinson JG. omega-3 fatty acids and domain-specific cognitive aging: secondary analyses of data from WHISCA. Neurology. 2013 Oct 22;81(17):1484-91. doi: 10.1212/WNL.0b013e3182a9584c. Epub 2013 Sep 25. PMID 24068783
- [Background] Goveas JS, Espeland MA, Hogan PE, Tindle HA, Shih RA, Kotchen JM, Robinson JG, Barnes DE, Resnick SM. Depressive Symptoms and Longitudinal Changes in Cognition: Women's Health Initiative Study of Cognitive Aging. J Geriatr Psychiatry Neurol. 2014 Jun;27(2):94-102. doi: 10.1177/0891988714522697. Epub 2014 Feb 28. PMID 24584465
- [Background] Driscoll I, Espeland MA, Wassertheil-Smoller S, Gaussoin SA, Ding J, Granek IA, Ockene JK, Phillips LS, Yaffe K, Resnick SM; Women's Health Initiative Study of Cognitive Aging. Weight change and cognitive function: findings from the Women's Health Initiative Study of Cognitive Aging. Obesity (Silver Spring). 2011 Aug;19(8):1595-600. doi: 10.1038/oby.2011.23. Epub 2011 Mar 10. PMID 21394095
- [Background] Resnick SM, Coker LH, Maki PM, Rapp SR, Espeland MA, Shumaker SA. The Women's Health Initiative Study of Cognitive Aging (WHISCA): a randomized clinical trial of the effects of hormone therapy on age-associated cognitive decline. Clin Trials. 2004;1(5):440-50. doi: 10.1191/1740774504cn040oa. PMID 16279282
- [Background] Espeland MA, Coker LH, Wallace R, Rapp SR, Resnick SM, Limacher M, Powell LH, Messina CR; Women's Health Initiative Study of Cognitive Aging. Association between alcohol intake and domain-specific cognitive function in older women. Neuroepidemiology. 2006;27(1):1-12. doi: 10.1159/000093532. Epub 2006 May 24. PMID 16717476
- [Background] Resnick SM, Maki PM, Rapp SR, Espeland MA, Brunner R, Coker LH, Granek IA, Hogan P, Ockene JK, Shumaker SA; Women's Health Initiative Study of Cognitive Aging Investigators. Effects of combination estrogen plus progestin hormone treatment on cognition and affect. J Clin Endocrinol Metab. 2006 May;91(5):1802-10. doi: 10.1210/jc.2005-2097. Epub 2006 Mar 7. PMID 16522699
- [Background] Resnick SM, Espeland MA, An Y, Maki PM, Coker LH, Jackson R, Stefanick ML, Wallace R, Rapp SR; Women's Health Initiative Study of Cognitive Aging Investigators. Effects of conjugated equine estrogens on cognition and affect in postmenopausal women with prior hysterectomy. J Clin Endocrinol Metab. 2009 Nov;94(11):4152-61. doi: 10.1210/jc.2009-1340. Epub 2009 Oct 22. PMID 19850684
- [Background] Espeland MA, Miller ME, Goveas JS, Hogan PE, Coker LH, Williamson J, Naughton M, Resnick SM; Whisca Study Group. Cognitive function and fine motor speed in older women with diabetes mellitus: results from the women's health initiative study of cognitive aging. J Womens Health (Larchmt). 2011 Oct;20(10):1435-43. doi: 10.1089/jwh.2011.2812. Epub 2011 Aug 5. PMID 21819251
- [Result] Espeland MA, Brunner RL, Hogan PE, Rapp SR, Coker LH, Legault C, Granek I, Resnick SM; Women's Health Initiative Study of Cognitive Aging Study Group. Long-term effects of conjugated equine estrogen therapies on domain-specific cognitive function: results from the Women's Health Initiative study of cognitive aging extension. J Am Geriatr Soc. 2010 Jul;58(7):1263-71. doi: 10.1111/j.1532-5415.2010.02953.x. PMID 20649689